CLINICAL TRIAL: NCT05456321
Title: tDCS and Cognitive Training as a Neurodevelopmental Intervention in FASD
Brief Title: CIFASD 5 tDCS and Cognitive Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSYCH-2022-30910
Record Dates: First submitted 2022-06-10; First posted 2022-07-13 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Fetal Alcohol Spectrum Disorders
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: 1:1 randomized allocation to active tDCS or placebo (sham tDCS).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and families will be blinded. The principal investigator will be blinded. The research staff member coordinating the visit will be blinded. The care provider is not involved in the research and is, therefore, blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cognitive Training and Active tDCS (Active Comparator): 5 sessions of computerized executive functioning training - plus active tDCS (also 5 sessions).
  Interventions: Device: Active tDCS; Behavioral: Cognitive Training
- Cognitive Training and Sham tDCS (Sham Comparator): 5 sessions of computerized executive functioning training - plus sham tDCS (also 5 sessions).
  Interventions: Behavioral: Cognitive Training; Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — Active Transcranial Direct Current Stimulation (tDCS)
  Arms: Cognitive Training and Active tDCS
Behavioral: Cognitive Training — Computerized Cognitive Training
Device: Sham tDCS — Sham Transcranial Direct Current Stimulation (tDCS)
  Arms: Cognitive Training and Sham tDCS

SUMMARY:
This is a randomized placebo-controlled trial of cognitive training with transcranial direct current stimulation (tDCS) for children and adolescents (ages 8 - 17 years) with prenatal alcohol exposure (PAE).

DETAILED DESCRIPTION:
Prenatal alcohol exposure (PAE) has profound detrimental effects on brain development and, as a result, has permanent consequences for cognition, learning, and behavior. Individuals with Fetal Alcohol Spectrum Disorders (FASD) commonly have a range of neurocognitive impairments that directly lead to practical problems with learning, attention, working memory, task planning/execution, and decision making, among other areas of functioning. Despite the profound public health burden posed by FASD, there have been very few treatment studies in this population. This study will examine the effects of a cognitive remediation training augmented with transcranial direct current stimulation (tDCS) in children and adolescents with PAE. The study involves a baseline visit with cognitive testing, 5 sessions of tDCS (including the baseline visit) with active and sham arms, a 6th visit for cognitive testing.

ELIGIBILITY:
Inclusion Criteria:

* Documented heavy prenatal alcohol exposure (self-report, social service records, or adoption records) and meeting criteria for an associated FASD diagnosis (FAS, partial FAS, or ARND).
* An available parent or legal guardian capable of giving informed consent

Exclusion Criteria:

* Substance abuse in the participant
* Neurological condition or other developmental disorder
* Serious psychiatric disorder known to affect brain functioning and cognitive performance Birthweight < 1500 grams
* MRI contraindication
* tDCS contraindication

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Continuous Performance Test performance | After each study visit (approx. bi-weekly) for the duration of the study (10 visits, approx. 5 weeks)
  Change in Continuous Performance Test performance
Change in Delis-Kaplan Executive Function System -Trail Making performance | Visit 1 and Visit 5 (approx. 3 weeks apart)
  Change in Delis-Kaplan Executive Function System - Trail Making performance
Change in Delis-Kaplan Executive Function System Color Word Interference performance | Visit 1 and Visit 5 (approx. 3 weeks apart)
  Change in Delis-Kaplan Executive Function System - Color Word Interference performance
Change in Wechsler Digit Span performance | Visit 1 and Visit 5 (approx. 3 weeks apart)
  Change in Wechsler Intelligence Scale for Children or Wechsler Adult Intelligence Digit Span performance
Change in Wechsler Picture Span performance | Visit 1 and Visit 5 (approx. 3 weeks apart)
  Change in Wechsler Intelligence Scale for Children or Wechsler Adult Intelligence Scale Picture Span performance

SECONDARY OUTCOMES:
Change in Oral Word Reading Fluency performance | Visit 1 and Visit 5 (approx. 3 weeks apart)
  Change in Oral Word Reading Fluency performance
Change in Math Fluency performance | Visit 1 and Visit 5 (approx. 3 weeks apart)
  Change in Mathematics Fluency performance

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Wozniak, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers.

DOCUMENTS (1):
  • Informed Consent Form (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/21/NCT05456321/ICF_000.pdf